CLINICAL TRIAL: NCT01291238
Title: Lifestyle Related Health and Health Promoting Activities for Youths With Intellectual Disabilities
Brief Title: School Intervention With Daily Physical Activity and Healthy Food for Students With an Intellectual Disability.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); City of Stockholm Competence Fund (Unknown); Lindeparkens upper secondary school for intellectual disability students (Unknown); Mälardalen University (Other); Health Care Sciences Postgraduate School at the Karolinska Institutet (Unknown)
Responsible Party: Claude Marcus, Karolinska Institutet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2009/772-32
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Weight Loss; Food Habits; Mental Retardation
Keywords: learning disability; blood lipids; cardio metabolic risk factors; upper secondary school for learning disability students; adolescents; cardio respiratory fitness; absorptiometry photos
MeSH Terms: conditions — Weight Loss; Feeding Behavior; Intellectual Disability; Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy lifestyle habits (Experimental): Increased physical activity and healthy food with decreased sugar and fat content
  Interventions: Behavioral: Healthier, Smarter, Happier

INTERVENTIONS:
Behavioral: Healthier, Smarter, Happier — Increased physical activity and decreased sugar and fat intake during school hours

SUMMARY:
A whole of school intervention with daily physical activity and healthy food for students with intellectual disabilities. The aim is to provide plenty of concrete examples of healthy life style choices and using school personnel and peers as role models. This will presumably result in healthier weight, better fitness and not least in new familiar healthy habits.

DETAILED DESCRIPTION:
Youth with an intellectual disability are reported more sedentary and more often overweight than non intellectual disability youth. Cardio metabolic risk factors are observed more frequent and at an earlier age among young people with intellectual disability. The school reaches all students and they spend the main part of their day in the school milieu hence examples of healthy lifestyle can be provided there.

This intervention increased physical activity with daily scheduled physical activity. At least one lesson each week was at the gym. Food provided in the school environment was considered from content of sugar and fat and ónly healthy food choices was available at school. This included all school activities, both in the school area and on school activities out in the community. It included home economic lessons as well as the school cafeterias supply and school lunch content.

To increase vegetable intake a special designed plate was used for lunch according the "plate model". In addition, the plate model was one theme during art class.

ELIGIBILITY:
Inclusion Criteria:

* mild/moderate intellectual disability
* students at the upper secondary schools for intellectual disability students

Exclusion Criteria:

* severe intellectual disability
* obesity related syndromes
* major physical disabilities

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 145 (Actual)
Dates: Start 2004-03; Primary Completion 2007-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Decrease in cardio metabolic risk factors | 2 years
  At baseline and after 2 years of intervention; height, weight, waist circumference, blood pressure was measured. In addition fasting blood samples of total cholesterol, triglycerides, fasting glucose and insulin. Absorptiometry photos (DXA) for body composition.
  Postintervention measures in addition compared to a controlgroup. Cross sectional data on all school students of all above mentioned variables and also cholesterol as HDL and LDL compared to a control group.

SECONDARY OUTCOMES:
Increase in physical fitness | 2 years
  At baseline and after 2 years of intervention a submaximal ergometer bicycle test. Postintervention measures in addition compared to a controlgroup.
  Cross sectional data on all school students from accelerometer, actiwatch, for frequency, intensity and level of physical activity compared to a control group.
Increased vegetable intake | at least 1 year
  To measure if the special plate made students take 37,5% vegetables or more as is the vegetable field on the plate.Effect of the specially designed plate according the plate-model evaluates in an observational study with videorecording and photos of a self served lunchportion on an ordinary plate in an experimental situation.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Marcus, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Department of clinical science, intervention and technology. Division of pediatrics, B62, Stockholm, Sweden